CLINICAL TRIAL: NCT03093519
Title: A Phase 1 Randomized, Double-blind, Placebo-controlled, Repeated Dose Study of KHK6640 in Japanese Patients With Alzheimer's Disease
Brief Title: A Repeated Dose Study of KHK6640 in Japanese Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6640-003
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KHK6640 (Experimental): Intravenous administration
  Interventions: Drug: KHK6640
- Placebo (Placebo Comparator): Intravenous administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KHK6640 — Intravenous administration
  Arms: KHK6640
Drug: Placebo — Intravenous administration
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of KHK6640, given as a repeated dose in Japanese patients with Mild to Moderate Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate Alzheimer's Disease
* Body weight ≥ 40 kg and < 100 kg
* Clinical Dementia Rating (CDR) score of 1 or 2
* Mini Mental State Examination (MMSE) score of ≥ 17 amd ≤ 26

Exclusion Criteria:

* Previous active treatment with an Alzheimer's Disease immunotherapy in an investigational study
* Use of another investigational drug within 16 weeks prior to the enrollment
* Subjects who meet National Institute of Neurological Disorders and Stroke/Association Internationale pour la Recherche et l'Enseignement en Neurosciences (NINDS/AIREN) criteria for vascular dementia
* Subjects with a history of presence of clinically significant seizures, brain trauma, transient ischemic attack, and/or cerebrovascular disease
* Subjects with a presence of a neurological condition that could be contributing to cognitive impairment above and beyond that caused by the subject's Alzheimer's Disease
* Subjects who have evidence of infection, tumor, or other clinically significant lesions that could indicate a dementia diagnosis other than Alzheimer's Disease

Ages: 55 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2017-12-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Up to 197days after first dosing
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- Closed information, Saitama, Japan

IPD SHARING:
Plan to Share IPD: No